CLINICAL TRIAL: NCT04537000
Title: Individualized Strategies of Red Blood Cell Transfusion for Perioperative Pediatric Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: transfusion-08-2020
Record Dates: First submitted 2020-08-25; First posted 2020-09-03 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-03

CONDITIONS: Individualized Transfusion Strategy; Red Blood Cell; Perioperative Pediatric Patient; Clinical Outcome
Keywords: transfusion; pediatric patient; individualized strategy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The strategies of red blood cell transfusion for the pediatric patients in this group will be made by the attending doctors in charge based on the current transfusion guidelines. The attending doctors decide when to start blood red cell transfusion and order the volume of the blood red cell as the usual clinical practice.
- study group (Experimental): For study group, the clinical condition score must be identified every time red blood cell transfusion is considered. The strategies of red blood cell transfusion for the pediatric patients in this group, including the trigger and the volume, will be made based on the comparison between the clinical condition score and the Hb concentration.
  Interventions: Diagnostic Test: clinical condition score

INTERVENTIONS:
Diagnostic Test: clinical condition score — A score is firstly identified using a clinical condition scale including the concentration of inspired oxygen to maintain the percutaneous oxygen saturation (SPO2)≧95%, the fusion rate of catecholamine drugs to maintain normal blood pressure, the nasopharyngeal temperature and the oxygen saturation of central venous blood. The score was graded as 0, 1 and 2 points according to the patient's clinical condition. The score identified from the scale plus 7 finally makes the clinical condition score. If the score is higher than 10, it will be replaced with 10. That is to say, the highest clinical condition score is 10. If the clinical condition score≦Hb, blood red cell transfusion will not be started. If the clinical condition score>Hb, blood red cell transfusion will be started, and the volume will be calculated using the following formulation, transfusion volume(ml)=(clinical condition score - Hb)*body weight *5.
  Arms: study group

SUMMARY:
The individualized strategies of red blood cell for perioperative pediatric patients are made based on the comparison between the clinical condition score and the Hb concentration.

DETAILED DESCRIPTION:
The hypothesis is that the individual transfusion strategies will help to save blood resource, and meanwhile will not adversely affect the patients' clinical outcomes. Participants will be randomly divided into two groups, where the strategies of transfusion of red blood cell will be made following different principles. The strategies for patients in control group will be made by the attending doctors in charge according to the current Chinese red blood cell transfusion guidelines. For the patients in study group, the clinical condition will be identified every time red blood cell transfusion is considered. The strategies will be made according to the comparison between the score and the Hb concentration. The volume of the red blood cell used in these two groups will be compared. The number of patients who need transfusion in these two groups will be compared. The clinical outcomes will also be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* The Hb concentration is tested before operation. It is higher than 7g/dl and lower than 10g/dl. Or it is anticipated that it will decrease lower than 10g/dl.

Exclusion Criteria:

* The patient will not undergo an operation.
* newborn or premature baby
* patients accompanied with hemorrhagic disease or cyanotic heart disease
* patients with ischemic heart disease or ischemic cerebrovascular disease

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
the volume of red blood cell (RBC) used adjusted to body weight | baseline through 3 days after surgery
  This is a repeated measurement data. The volume of RBC used adjusted to body weight = the volume of RBC (ml) used/ body weight(Kg). It is repeatedly recorded during this time frame. The data for intraoperation phase, for postoperation phase and for both intraoperation and postoperation phase are analyzed.The data would be measured at baseline (before operation), at the end of operation and on the 3rd days after operation.

SECONDARY OUTCOMES:
hemoglobin （Hb） concentration | baseline through 3 days after surgery
  Hb concentration is assessed by blood gas test. It is a repeated measurement data.
heart rate | during operation(about 2-6 hours)
  It is a repeated measurement data. It is recorded every 5-10 minutes during this time frame .
blood pressure（Systolic） | during operation (about 2-6 hours)
  It is a repeated measurement data. It is (Systolic blood pressure ) recorded every 5-10 minutes during this time frame .
blood pressure（Diastolic） | during operation (about 2-6 hours)
  It is a repeated measurement data. It is ( Diastolic blood pressure ) recorded every 5-10 minutes during this time frame .
lactate (Lac) | during operation (about 2-6 hours)
  It is a repeated measurement data. It is recorded every time blood gas test is ordered during this time frame.
length of stay in post anesthesia care unit (PACU) | about 2-6 hours
  the time between the arrival of the patient to the PACU to the discharge to the ward
infection | from the end of operation to the 3rd month after the operation.
  It is a binary variable. The data will be set as "1" if the patients got any infections such as wound infection, sepsis, etc. It will be set as "0" if there is no evidence for infection.
unexpected transfer to intense care unit (ICU) | from the end of operation to the 3rd day after the operation.
  It is a binary variable. The data will be set as "1" if the patient is transferred to ICU unexpectedly. It will set as "0" if not.
length of stay in hospital after operation | from the date of operation to discharge （about 1-4 weeks ）
  from the date of the operation to the date when the patient is discharged
the number of patients who need RBC transfusion | baseline through 3 days after surgery
  This is a repeated measurement data. The number of patients who need RBC transfusion during operation and during the first 3 days after operation is recorded, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Shi, Master, Study Chair — Children's Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavoie J. Blood transfusion risks and alternative strategies in pediatric patients. Paediatr Anaesth. 2011 Jan;21(1):14-24. doi: 10.1111/j.1460-9592.2010.03470.x. PMID 21155923
- [Background] Carson JL, Carless PA, Hebert PC. Transfusion thresholds and other strategies for guiding allogeneic red blood cell transfusion. Cochrane Database Syst Rev. 2012 Apr 18;4(4):CD002042. doi: 10.1002/14651858.CD002042.pub3. PMID 22513904
- [Background] AABB white papers: building a better patient blood management program identifying tools, soving problems and promoting patient safety; 2015
- [Background] Carson JL, Guyatt G, Heddle NM, Grossman BJ, Cohn CS, Fung MK, Gernsheimer T, Holcomb JB, Kaplan LJ, Katz LM, Peterson N, Ramsey G, Rao SV, Roback JD, Shander A, Tobian AA. Clinical Practice Guidelines From the AABB: Red Blood Cell Transfusion Thresholds and Storage. JAMA. 2016 Nov 15;316(19):2025-2035. doi: 10.1001/jama.2016.9185. PMID 27732721
- [Background] Kozek-Langenecker SA, Ahmed AB, Afshari A, Albaladejo P, Aldecoa C, Barauskas G, De Robertis E, Faraoni D, Filipescu DC, Fries D, Haas T, Jacob M, Lance MD, Pitarch JVL, Mallett S, Meier J, Molnar ZL, Rahe-Meyer N, Samama CM, Stensballe J, Van der Linden PJF, Wikkelso AJ, Wouters P, Wyffels P, Zacharowski K. Management of severe perioperative bleeding: guidelines from the European Society of Anaesthesiology: First update 2016. Eur J Anaesthesiol. 2017 Jun;34(6):332-395. doi: 10.1097/EJA.0000000000000630. PMID 28459785
- [Background] Rouette J, Trottier H, Ducruet T, Beaunoyer M, Lacroix J, Tucci M; Canadian Critical Care Trials Group; PALISI Network. Red blood cell transfusion threshold in postsurgical pediatric intensive care patients: a randomized clinical trial. Ann Surg. 2010 Mar;251(3):421-7. doi: 10.1097/SLA.0b013e3181c5dc2e. PMID 20118780
- [Background] Zhang F, Zheng ZB, Zhu ZQ, Liu DX, Liu J. Application of Perioperative Transfusion Trigger Score in Patients Undergoing Surgical Treatment of Malignant Tumor. Indian J Hematol Blood Transfus. 2020 Jan;36(1):156-163. doi: 10.1007/s12288-019-01180-z. Epub 2019 Sep 12. PMID 32158099
- [Background] New HV, Grant-Casey J, Lowe D, Kelleher A, Hennem S, Stanworth SJ. Red blood cell transfusion practice in children: current status and areas for improvement? A study of the use of red blood cell transfusions in children and infants. Transfusion. 2014 Jan;54(1):119-27. doi: 10.1111/trf.12313. Epub 2013 Jun 30. PMID 23808415